CLINICAL TRIAL: NCT04777487
Title: Evaluation of Peptidyl Arginine Deiminase 4 (PAD4), Galectin-3 and TNF-α Levels in Gingival Crevicular Fluid of Patients With Different Periodontal Diseases
Brief Title: Evaluation of Biomarker Levels in Gingival Crevicular Fluid of Patients With Different Periodontal Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Hazal Akkaya, Research Assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-TDU-DİŞF-0008
Record Dates: First submitted 2021-02-27; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) samples of GCF were obtained from 60 systemically healthy non-smoker individuals with periodontitis (P, n=20), gingivitis(G, n=20) and healthy periodontium (S, n=20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Periodontium (Experimental): Full-mouth clinical periodontal measurements recorded and GCF obtained.
  Interventions: Diagnostic Test: GCF obtaining
- Gingivitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF obtained.
  Interventions: Diagnostic Test: GCF obtaining
- Periodontitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF obtained.
  Interventions: Diagnostic Test: GCF obtaining

INTERVENTIONS:
Diagnostic Test: GCF obtaining — 4 samples of gingival crevicular fluid, 1 from each quadrant of the patient's jaw, were collected by means of paper strips.

SUMMARY:
Objectives: The aim of this study is; detection of peptidyl arginine deiminase4 (PAD4), galectin-3 and tumor necrosis factor alpha (TNF-α) levels in gingival crevicular fluid (GCF) samples of periodontally healthy, gingivitis and periodontitis patients and the possible correlation between these values and clinical parameters of periodontal diseases. Materials and methods: Samples of GCF were obtained from 60systemically healthy non-smoker individuals with periodontitis (P, n=20), gingivitis(G, n=20) and healthy periodontium (S, n=20). Full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were also recorded. Enzyme-linked immunosorbent assay (ELISA) was used to determine PAD4, galectin-3 and TNF-α levels in the biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (The determination of healthy volunteers will be based on the statements of the patients in the anamnesis. No additional examinations will be made.)
* At least twenty permanent teeth in the mouth
* Non-smoker
* No medication for continuous use
* Those who have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months.
* Not in pregnancy or lactation period.
* For the periodontitis group that has not received periodontal treatment in the last 6 months
* For the periodontitis group; According to the evaluation made in 6 regions of each tooth, individuals with 30% or more bleeding on probing area, at least 2 teeth not adjacent to each quarter jaw with a depth of 5 mm or more and 4 mm or more attachment loss, coronal 1/3 and more on radiography (horizontal and / or vertical) bone loss
* For the gingivitis group; According to the evaluation made in 6 regions of each tooth, individuals with 10% or more bleeding on probing area, having a probing depth of less than 4mm and no attachment loss
* For healthy group; According to the evaluation made in 6 regions of each tooth,individuals with less than 10% bleeding on probing area, having a probing depth less than 4mm and no loss of attachment were included in the study.

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months
* Smokers are not included in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
The total amount of Galectin-3 in GCF | 24 hours after taking the clinical measurements at the first visit
  The total amount of Galectin-3 in GCF
The total amount of PAD4 in GCF | 24 hours after taking the clinical measurements at the first visit
  The total amount of PAD4 in GCF

SECONDARY OUTCOMES:
The total amount of TNF-α in GCF | 24 hours after taking the clinical measurements at the first visit
  The total amount of TNF-α in GCF

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sağlam, Study Director — Izmir Katip Çelebi University
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF